CLINICAL TRIAL: NCT02341118
Title: Capturing BRCA1/2 Mutational Status in Women With High Grade Serous Ovarian Cancer and Impact on Clinical Outcome.
Status: Terminated | Type: Observational
Why Stopped: This study did not collect sufficient data for primary endpoint analysis.
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: BRCA Screening
Record Dates: First submitted 2014-11-27; First posted 2015-01-19 (Estimated); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Ovarian Cancer
Keywords: BRCA1/2 Mutational Status
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Genetic: BRCA genetic data — Two blood samples will be taken which is part of the standard of care. Tumor samples will be obtained from previous biopsy or surgery prior to this study for DNA testing

SUMMARY:
BRCA1 or BRCA2 genes, are implicated in 10-15% of ovarian cancer cases, increased to 22% germline BRCA1/2 mutation frequency in patients with high grade serous histology subtype, including those women who have no family history of breast or ovarian cancer. With the rapid advancement of therapeutics targeted this population, this protocol seeks to provide genetic BRCA1/2 screening to all patients with high grade serous ovarian cancer. This information may help in selection of future treatment options and genetic testing for BRCA1/2 may be used to potentially prevent a proportion of cancer for the family members.

This study will be an opportunity for patient to improve access at genetic and molecular testing for BRCA1/2 mutation which could impact her future treatment option. Moreover, this study will allow to prospectively assess the proportion of patients with BRCA mutation in ovarian cancer and describe the type of mutations identified in a large population.

DETAILED DESCRIPTION:
Primary Objectives

· To provide genomic profiling for BRCA1 and BRCA2 mutational status in patients' with high grade serous ovarian cancer.

Secondary Objectives

* To track the number of women with high grade serous ovarian cancer who are being screened in Princess Margaret Cancer Center for mutations in BRCA1/2
* To track accrual rates and clinical outcomes in patients with high grade serous ovarian cancer who are BRCA1/2-positive
* To correlate impact of BRCA1/2 mutational status on clinical outcome
* To track utilization of genetic counseling services at Princess Margaret Cancer Centre

ELIGIBILITY:
Inclusion Criteria:

* Patients with high grade serous carcinoma originating from the ovaries, fallopian tube or peritoneal cavity; subtype of high grade endometrioid and clear cell ovarian cancer could be eligible in the exploratory cohort
* Patient must be ≥18 years old
* All patients must have sufficient archival tumor tissue for molecular analysis
* All patients must consent to have a genetic testing
* All patients must have signed and dated an informed consent form

Exclusion Criteria:

· Other histology subtype

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with high grade serous carcinoma originating from the ovaries, fallopian tube or peritoneal cavity; subtype of high grade endometrioid and clear cell ovarian cancer could be eligible in the exploratory cohort
Sampling Method: Non-Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2014-05; Primary Completion 2018-04 (Actual); Study Completion 2023-05-08 (Actual)

PRIMARY OUTCOMES:
genomic profiling for BRCA1 and BRCA2 mutational status in patients' with high grade serous ovarian cancer. | upon availability of genetic consultation report min 6 weeks
  participants will also be followed for all treatments and responses until death

CONTACTS AND LOCATIONS:
Overall Officials: Amit Oza, Principal Investigator — University Health Network, Toronto
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada